CLINICAL TRIAL: NCT06825260
Title: Polyethylene Glycol 3350 Compared With Senna After Urogynecologic Surgery A Randomized Controlled Trial
Brief Title: PEG3350 vs Senna After Urogyn Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Health, New York (Other)
Responsible Party: Principal Investigator, Keila S. Muniz, MD, Physician, St. Joseph's Physicians Urogynecology, St. Joseph's Health, New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StJosephNewYork
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Defecation Syndrome; Postoperative Constipation
Keywords: obstructive defecation syndrome (ODS); Postoperative constipation
MeSH Terms: interventions — Sennosides; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Senna (Experimental): Senna (Sennosides), oral, 8.6mg, 2 tablets daily (up to 4 tablets twice a day) for 7 days
  Interventions: Drug: Senna
- Polyethylene Glycol 3350 (Active Comparator): Polyethylene Glycol 3350, oral, 17g, daily for 7 days
  Interventions: Drug: Polyethylene glycol 3350

INTERVENTIONS:
Drug: Senna — Senna, oral, 8.6mg, 2 tablets daily (up to 4 tablets twice a day) for 7 days
  Other Names: Senokot; Sennoside
  Arms: Senna
Drug: Polyethylene glycol 3350 — Polyethylene Glycol 3350, oral, 17g, daily for 7 days
  Other Names: PEG 3350; Miralax
  Arms: Polyethylene Glycol 3350

SUMMARY:
The goal of this study is to evaluate whether polyethylene glycol 3350 (PEG3350) versus senna is better at relieving postoperative constipation after urogynecologic surgery. The main questions it aims to answer are:

What number of patients taking PEG3350 have obstructed defecation syndrome (ODS), a form of constipation, vs those taking senna in the week after urogynecologic surgery? What patient-level and procedure-level characteristics are associated with postoperative ODS, in patients taking PEG3350 vs senna? participants will: Take their randomized medication daily for seven days after surgery Fill out an ODS questionnaire before and one week after surgery Complete a daily bowel diary for 7 days after surgery

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether polyethylene glycol 3350 (PEG3350) versus senna is superior in the setting of postoperative constipation after urogynecologic surgery. This is a randomized controlled trial with the aim of comparing PEG3350 vs senna as postoperative recommended treatment for obstructive defecation constipation. Our hypothesis is that senna decreases the proportion of women with obstructive defecation constipation compared to use of PEG3350 after urogynecologic surgery. Women 18 years of age and older undergoing surgery for pelvic organ prolapse, stress urinary incontinence or both by the Department of Urogynecology at St. Joseph's Health Hospital, will be randomized to one of two study arms: senna or PEG3350. Arm 1: Polyethylene Glycol 3350, 17g, daily, oral. Arm 2: Senna (Sennosides) 8.6mg, 2 tablets daily, oral (up to 4 tablets twice a day). Interventions would be administered after surgery on postoperative day #0 and continue for 7 days total.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes women scheduled for urogynecologic surgery for pelvic organ prolapse and/or stress urinary incontinence and at least 18 years old.

Exclusion Criteria:

* Exclusion criteria include undergoing concomitant bowel surgery (colonic resection, anal sphincter repair, rectovaginal fistula repair, rectopexy) or placement of a sacral neuromodulation device alone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative ODS in Patients Taking PEG3350 vs Senna | From enrollment to the end of treatment at 7 days after surgery.
  The primary outcome is to determine the proportion of patients with postoperative obstructed defecation syndrome (ODS), defined as a score of nine or greater on the ODS questionnaire, in patients taking PEG3350 vs senna in the week after urogynecologic surgery.

SECONDARY OUTCOMES:
Patient-level and Procedure-level Characteristics associated with Postoperative ODS in Patients Taking PEG3350 vs Senna | From enrollment to the end of treatment at 7 days after surgery.
  In order to identify postoperative bowel symptoms associated with ODS, enrolled participants will complete a bowel diary for 7 days after surgery. The bowel diary will include: type of bowel movement using the validated Bristol stool scale, degree of strain and pain measured on an 11-point numerical rating scale from 0-10 (zero denoting no presence of symptom and ten denoting the most severe symptom experienced), presence of splinting with bowel movements, sensation of incomplete evacuation (measured on an 11-point numerical rating scale from 0-10), additional medications taken to assist with bowel movements, fecal urgency, fecal incontinence, narcotic medication usage as well as time to first bowel movement. ODS score will be obtained preoperatively. Participants will be asked to estimate their preoperative frequency of bowel movements. Patients will self-identify their racial background. Medical records will be reviewed to obtain patient characteristics and perioperative data.

CONTACTS AND LOCATIONS:
Overall Officials: Keila S Muniz, MD, Principal Investigator — St. Joseph's Health
Locations (1):
- St. Joseph's Health Hospital, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No